CLINICAL TRIAL: NCT01205880
Title: Spray® and Vectical Ointment® in the Treatment of Plaque Psoriasis
Brief Title: Study to Evaluate Vectical in Combination With Clobex Spray to Treatment Plaque Psoriasis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Emer, Jason, M.D. (Individual)
Collaborators: Galderma Laboratories (Other)
Responsible Party: Jason Emer, M.D., Mount Sinai School of Medicine
Allocation: Randomized | Masking: Single | Purpose: Treatment
Other Study IDs: 08-1500
Record Dates: First submitted 2010-09-17; First posted 2010-09-21 (Estimated); Last update posted 2010-09-21 (Estimated); Status verified 2010-09

CONDITIONS: Psoriasis
Keywords: combination treatment; topical corticosteroid; vitamin D analogue; clobex; vectical; clobetasol; calcitriol
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- vectical ointment and clobex spray (Active Comparator): patients were assigned to apply vectical ointment first then clobex spray on one target lesion and also apply clobex spray first then vectical ointment on a different target lesion on the opposite side of the body.
  Interventions: Drug: Calcitriol ointment; Drug: Clobetasol spray

INTERVENTIONS:
Drug: Calcitriol ointment — twice daily
  Other Names: Vectical Ointment
Drug: Clobetasol spray — twice daily
  Other Names: Clobex spray

SUMMARY:
This investigator-blinded study is designed to assess whether the order of application affects the efficacy of the combination treatment Clobex® Spray (clobetasol propionate) and Vecitcal® (calcitriol) Ointment in plaque psoriasis.

DETAILED DESCRIPTION:
This is an investigator-blinded, bilateral comparison study. A total of up to 12 subjects with mild to moderate plaque psoriasis will be enrolled in this study, so that at least 10 subjects complete the 4 week trial. These 12 subjects will receive the combination therapy of Clobex® Spray and Vectical® Ointment to treat their psoriatic lesions (except those on the scalp, face, groin, axillae or other intertriginous areas). Half of the subjects will first apply the Clobex® Spray followed by the Vectical ointment to lesions on the right side of their bodies, and Vectical® Ointment first followed by Clobex® Spray to the lesions of the left side of their bodies. The other half of the subjects will first apply Clobex® Spray followed by Vectical® Ointment to the lesions of the left side of their bodies, and Vectical® Ointment first followed by Clobex® Spray to the lesions on right side of their bodies. Treatment will be applied twice daily for 4 weeks. One target area on each side of the subject's body will be chosen for target lesion assessment.

All subjects will be consented prior to any study evaluations/procedures. Study evaluations including Target Lesion Severity Score (TLSS) and photography will be performed at Baseline/Day 0, week 2 and week 4.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be at least 18 years of age and in good general health as confirmed by a medical history.
2. Females of childbearing potential must have a negative urine pregnancy test on Baseline/Day 0 and must agree to use adequate birth control methods during the entire study (a barrier method {condoms, diaphragm}; hormonal contraceptives {birth control pills, implants [Norplant] or injections [DepoProvera]}; intrauterine device {IUD}; or abstinence {no sexual activity}).
3. Subjects must be diagnosed with plaque psoriasis affecting < 20% body surface area, with at least one discreet plaque on the each side of the body (excluding the face, scalp, groin, axillae or other intertriginous areas).
4. Subjects must have at least 2 lesions suitable for evaluating response to test agents (one on the right side and one on the left side of the body). The severity of the disease for each target lesion at Baseline/Day 0 must be rated at least 2 (Mild) for each of the key psoriasis characteristics (scaling, erythema, and plaque elevation).
5. Subjects must be able to understand the requirements of the study abide by the restrictions and return for the required examinations.

Exclusion Criteria:

1. Female subjects who are pregnant, nursing or planning a pregnancy during the study.
2. Subjects with known hypersensitivity to any components of the test medication.
3. Subjects with non-plaque psoriasis (e.g. guttate, erythrodermic) or other related diseases not classified as plaque psoriasis.
4. Subjects whose psoriasis involves only the scalp, face, groin, axillae, and/or other intertriginous areas.
5. Subjects who have surface area involvement too large (>20% BSA) that would require more than 59 ml/week (50 g/week) of Clobex® spray and/or more than 200 g/week of Vectical® ointment.
6. Subjects requiring any other medication (topical or systemic) that may affect the course of the disease during the study period as determined by the study investigators.
7. Subjects using biologics or any other systemic treatment (e.g. immunosuppressants, acitretin) for psoriasis within 12 weeks of entering the study.
8. Subjects using systemic corticosteroids within 28 days of entering the study
9. Subjects using topical corticosteroids or other topical therapies (other than emollients) at the target area locations within 2 weeks of entering the study
10. Subjects using phototherapy (UVB, PUVA) within 4 weeks of entering the study.
11. Subjects with overt pre-existing telangiectasias or skin atrophy at intended treatment sites (target areas).
12. Subjects with intakes of more than 2,000 IU/day (50 mcg/day) of vitamin D (tolerable upper intake level) and/or more than 1,000 mg/day of calcium (based on Dietary Reference Intakes developed by the Institute of Medicine of the National Academy of Sciences).
13. Subjects who have participated in another investigational drug or device research study (at the target areas) within 30 days of enrollment.
14. Subjects who are using any medication or has any disease which in the judgment of the investigator will interfere with the conduct or interpretation of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2009-12; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
improvement in target lesion severity score (TLSS) | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jason J Emer, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai School of Medicine, New York, New York, United States

REFERENCES:
- [Background] Jarratt MT, Clark SD, Savin RC, Swinyer LJ, Safley CF, Brodell RT, Yu K. Evaluation of the efficacy and safety of clobetasol propionate spray in the treatment of plaque-type psoriasis. Cutis. 2006 Nov;78(5):348-54. PMID 17186795
- [Background] Beutner K, Chakrabarty A, Lemke S, Yu K. An intra-individual randomized safety and efficacy comparison of clobetasol propionate 0.05% spray and its vehicle in the treatment of plaque psoriasis. J Drugs Dermatol. 2006 Apr;5(4):357-60. PMID 16673804
- [Background] Menter A, Korman NJ, Elmets CA, Feldman SR, Gelfand JM, Gordon KB, Gottlieb A, Koo JY, Lebwohl M, Lim HW, Van Voorhees AS, Beutner KR, Bhushan R; American Academy of Dermatology. Guidelines of care for the management of psoriasis and psoriatic arthritis. Section 3. Guidelines of care for the management and treatment of psoriasis with topical therapies. J Am Acad Dermatol. 2009 Apr;60(4):643-59. doi: 10.1016/j.jaad.2008.12.032. Epub 2009 Feb 13. PMID 19217694
- [Background] Abramovits W. Calcitriol 3 microg/g ointment: an effective and safe addition to the armamentarium in topical psoriasis therapy. J Drugs Dermatol. 2009 Aug;8(8 Suppl):s17-22. PMID 19702032
- [Background] Bruner CR, Feldman SR, Ventrapragada M, Fleischer AB Jr. A systematic review of adverse effects associated with topical treatments for psoriasis. Dermatol Online J. 2003 Feb;9(1):2. PMID 12639460